CLINICAL TRIAL: NCT03271255
Title: Apatinib Versus Bevacizumab in Combination With Second-line FOLFIRI in Patients With Metastatic Colorectal Cancer That Progressed During or After First-line Bevacizumab Plus an Oxaliplatin-based Regimen: A Randomised Phase 2 Trial
Brief Title: Apatinib Versus Bevacizumab in Second-line Therapy for Colorectal Cancer(ABST-C)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shenzhen People's Hospital (Other)
Responsible Party: Principal Investigator, Ruilian Xu, Dean of Oncology Department, Shenzhen People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Shenzhen CRC-001
Record Dates: First submitted 2017-08-31; First posted 2017-09-05 (Actual); Last update posted 2019-01-23 (Actual); Status verified 2018-12

CONDITIONS: Colorectal Neoplasms; Intestinal Neoplasms; Gastrointestinal Neoplasms; Digestive System Neoplasms
Keywords: apatinib; bevacizumab; FOLFIRI; colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Intestinal Neoplasms; Gastrointestinal Neoplasms; Digestive System Neoplasms | interventions — apatinib; Bevacizumab

STUDY DESIGN:
Intervention Model Description: Head-to-head comparison of apatinib versus bevacizumab plus sencond-line chemotherapy regimen FOLFIRI for treatment of metastatic colorectal cancer
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm Apatinib (Experimental): Apatinib-FOLFIRI:
  Apatinib Mesylate Tablets 500 mg po qd; Irinotecan 180 mg/m2 IV over 30-90 minutes,day 1; Leucovorin 400 mg/m2 IV infusion to match duration of irinotecan infusion,day 1; 5-FU 400 mg/m2 IV bolus day 1,then 1200 mg/m2/d x 2 days (total 2400 mg/m2 over 46-48 hours) continuous infusion; Repeat every 2 weeks.
  Interventions: Drug: Apatinib Mesylate Tablets
- Arm Bevacizumab (Active Comparator): Bevacizumab-FOLFIRI:
  Bevacizumab Injection 5 mg/kg IV over 30 minutes,day 1; Irinotecan 180 mg/m2 IV over 30-90 minutes,day 1; Leucovorin 400 mg/m2 IV infusion to match duration of irinotecan infusion,day 1; 5-FU 400 mg/m2 IV bolus day 1,then 1200 mg/m2/d x 2 days (total 2400 mg/m2 over 46-48 hours) continuous infusion; Repeat every 2 weeks.
  Interventions: Drug: Bevacizumab Injection

INTERVENTIONS:
Drug: Apatinib Mesylate Tablets — Apatinib combination with FOLFIRI regimen as the second-line chemotherapy for mCRC
  Other Names: YN968D1
  Arms: Arm Apatinib
Drug: Bevacizumab Injection — Bevacizumab combination with FOLFIRI regimen as the second-line chemotherapy for mCRC
  Other Names: Avastin
  Arms: Arm Bevacizumab

SUMMARY:
Bevacizumab, as an antibody of vascular endothelial generated factor (VEGF), combined with the fluorouracil-based chemotherapy regimens for metastatic colorectal cancer, has become the classical first-line treatment. However, vast majority of patients eventually will suffer progression disease. The second-line treatment includes replacing chemotherapy regimens whistle continuing bevacizumab or other anti-VEGF antibodies, such as Aflibercept and Ramucirumab. Apatinib is a small molecule tyrosine kinase inhibitor (TKI), which can highly selectively bind to and strongly block VEGF receptor 2 (VEGFR - 2), also potently suppress the activities of Ret, c-kit and c-src, resulting in reduced cell migration, proliferation, and tumor microvascular density mediated by VEGF .There are already robust data showing that antibodies aimed at blocking VEGF signaling pathways combined with chemotherapy to treat advanced colorectal cancer is superior as compared to chemotherapy alone. Thus, we hypothesize that the effect of using the second-line chemotherapy regimens combined with apatinib may be superior to those combined with bevacizumab. In this study,the patients who have progressed following or on first-line oxaliplatin and 5-FU combined with bevacizumab are randomised into two arms. Patients in the experimental arm receive second-line FOLFIRI combined with apatinib and those in the control arm receive second-line FOLFIRI combined with bevacizumab. To compare the efficacy and safety of the two arms, progression-free survival(PFS) is the primary end point.If apatinib is superior to bevacizumab in the second-line setting,it is one possible option of anti-angiogenic therapy in combination with second-line FOLFIRI for treatment of advanced colorectal cancer.

DETAILED DESCRIPTION:
Firstly, screen eligible mCRC patients for enrolment. Our CRC clinical nurse specialists will document medical history of patients including diagnoses, first-line chemotherapy (mFOLFOX6 or CAPOX),bevacizumab dosage,toxicities,PFS on previous therapy.In the meantime,chest-abdonimal-pelvic CT and blood tests are to be examined to assess base-line measurable lesions and guarantee adequate organ function prior to enrolment.If all the values meet the criteria for enrolment, consent will be signed.

Secondly, randomise patients into two arms: Arm A-apatinib plus FOLFIRI regimen and arm B-bevacizumab plus FOLFIRI regimen.A software which is alike the procedure of coin flipping is used to randomise eligible patients.According to the selected regimen in specific arm,patients will be given full-dose drugs or reduced dose drugs if serious toxicities ( CTCAE v4.0 criteria grade 3/4) are complained since previous cycle of treatment.Symptoms and blood test results (including CEA and CA199) before each cycle will be recorded and the consultant oncologist, who is responsible for individual participants, will decide whether to continue next cycle chemotherapy with apatinib or bevacizumab based on the assigned arm.Radiological assessment consisting of chest-abdonimal-pelvic CT will be performed every 2 months.Notably,the monitor will check with physicians and nurse specialists for the accuracy and completeness of all data.

Thirdly, follow up participants and analyse primary end point (PFS) and secondary end points (OS,ORR and DCR).The causes of confirmed missing data in the trial should be recorded in detail to determine the mechanism of missing data and choose the suitable missing data handling methods.

ELIGIBILITY:
Inclusion Criteria:

* Inoperable colorectal adenocarcinoma excluding vermiform appendix cancer and anal canal cancer confirmed by histology
* Age ≥18 years ≤ 70 years at the time of informed consent
* ECOG performance status (PS) ≤ 1
* Provided informed consent before study-specific screening procedures
* Life expectancy not less than 90 days
* Participants have progressive disease on or within 6 months post the combination of bevacizumab and FOLFOX or CAPOX as the first-line chemotherapy for metastatic colorectal cancer
* Adequate organ function based on the following laboratory values obtained within 14 days prior to enrolment (excluding patients who received blood transfusions or hematopoietic growth factors within 14 days before the laboratory test) Neutrophil count: ≥1500/mm3 Platelet count: ≥10.0 x 104/mm3 Hemoglobin: ≥9.0 g/dL Total bilirubin: ≤1.5 mg/dL AST, ALT: ≤100 IU/L (≤200 IU/I if liver metastases present) Serum creatinine: ≤1.5 mg/dL Measurable or nonmeasurable disease based on the Response Evaluation Criteria in Solid Tumors, Version 1.1 (RECIST v1.1)
* Adequate blood coagulation function [International Normalized Ratio (INR) ≤1.5 and Partial Thromboplastin Time (PTT) or activated PTT (aPTT) ≤1.5 x upper limit of normal (ULN)). Participants on full-dose anticoagulation must be in a stable phase of anticoagulant therapy and if taking oral anticoagulation, participants must have an INR ≤3 without clinically significant active bleeding or a high risk of bleeding
* A historical colorectal cancer tissue sample is available for assessment of biomarkers with signed consent
* Signed informed consent to be provided

Exclusion Criteria:

* History of other malignancy with a disease-free survival <5 years (excluding curatively treated cutaneous basal cell carcinoma, curatively treated cervical in situ carcinoma , and gastroenterological carcinoma confirmed to be cured by endoscopic mucosal resection)
* With a large amount of pleural effusions or ascites requiring intervention
* Radiological evidence of brain metastases or brain tumor
* Actively infectious condition including hepatitis
* One of the following complications: 1) Gastrointestinal obstruction (including paralytic ileus) or gastrointestinal bleeding 2) Symptomatic cardiac disease (including unstable angina, myocardial infarction, and heart failure) 3) Pulmonary fibrosis or interstitial pneumonia 4) Uncontrolled diarrhea (that affects daily activities although adequate therapy 5) Uncontrolled diabetes mellitus
* One of the following medical histories: 1) Myocardial infarction: One episode within one year prior to enrollment or two or more lifetime episodes 2) Remarkable hypersensitivity to any of the study drugs ii) History of side effect to fluoropyrimidines suggestive of dihydropyrimidine dehydrogenase (DPD) deficiency
* Pregnant or lactating females, and males and females reluctant to use contraception
* Psychiatric disability that would disturb study compliance
* Other conditions determined by the investigator to be not suitable for participation in the study
* History of concurrent gastrointestinal perforation or gastrointestinal perforation within 1 year prior to enrollment
* Pulmonary hemorrhage/hemoptysis ≥ Grade 2 (identified as bright red blood of not less 2.5mL) within 1 month before enrollment.
* History of thoracotomy,laparotomy, or intestinal resection within 28 days prior to enrollment
* Unhealed wound (other than suture wounds due to implantation of a central venous port), traumatic fracture, or gastrointestinal ulcer
* Current cerebrovascular disease or thromboembolism or either within 1 year before enrollment
* Current anticoagulation therapy or requiring anticoagulation agents (> 325 mg/day of aspirin)
* Bleeding diathesis, coagulopathy, or coagulation factor abnormality (INR ≥1.5 within 14 days before enrollment)
* Uncontrolled hypertension Urine dipstick for proteinuria >+2

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-05-23 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival (PFS) Time | The follow-up period ranges from the first patient recruited to the last patient within 6 months after admission, up to 2 years
  PFS was defined as the time from the date of randomization until the date of objectively determined progressive disease (PD) [according to Response Evaluation Criteria in Solid Tumors (RECIST) version (v). 1.1] or death due to any cause, whichever was first. PD is at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 millimeters (mm). Participants who died without a reported prior progression were considered to have progressed on the day of their death. Participants who did not progress or were lost to follow-up were censored at the day of their last radiographic tumor assessment.

SECONDARY OUTCOMES:
Overall Survival (OS) | The follow-up period ranges from the first patient recruited to the last patient within 6 months after admission,up to 2 years
  OS was defined as the time in months from the date of randomization to the date of death from any cause. For participants not known to have died as of the cut-off date, OS was censored at the last known date alive.
Percentage of Participants Achieving an Objective Response (Objective Response Rate) | The follow-up period ranges from the first patient recruited to the last patient within 3 months after admission.
  The objective response rate is equal to the proportion of participants achieving a best overall response of partial response or complete response (PR + CR). Response was defined using RECIST, v. 1.1 criteria. CR was defined as the disappearance of all target and non-target lesions and any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm and normalization of tumor marker level of non-target lesions; PR was defined as having at least a 30% decrease in sum of longest diameter of target lesions taking as reference the baseline sum diameter.
Percentage of Participants Achieving a Stable Disease (SD) or a confirmed CR or PR (Disease Control Rate) | The follow-up period ranges from the first patient recruited to the last patient within 3 months after admission.
  Participants achieved disease control if they had a best overall response of CR, PR or SD. According to RECIST v1.1, CR was the disappearance of all non-nodal target lesions, with the short axes of any target lymph node reduced to <10 mm, the disappearance of all non-target lesions, and the normalization of tumor marker levels (if tumor markers were initially above the ULN); PR was defined as at least a 30% decrease in the sum of the diameters of target lesions (including the short axes of any target lymph node), taking as reference the baseline sum diameter. SD was neither sufficient shrinkage to qualify as PR nor sufficient increase to qualify as PD, taking as reference the smallest sum diameter since treatment started.

CONTACTS AND LOCATIONS:
Overall Officials: Ruilian Xu, MD, Principal Investigator — Shen Zhen People's Hospital
Locations (1):
- Shenzhen People's Hospital, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
All data will be shared with other researchers.
Supporting Information: Study Protocol, CSR
Time Frame: After the data is formally published.
Access Criteria: Open access.

REFERENCES:
- [Background] Bennouna J, Sastre J, Arnold D, Osterlund P, Greil R, Van Cutsem E, von Moos R, Vieitez JM, Bouche O, Borg C, Steffens CC, Alonso-Orduna V, Schlichting C, Reyes-Rivera I, Bendahmane B, Andre T, Kubicka S; ML18147 Study Investigators. Continuation of bevacizumab after first progression in metastatic colorectal cancer (ML18147): a randomised phase 3 trial. Lancet Oncol. 2013 Jan;14(1):29-37. doi: 10.1016/S1470-2045(12)70477-1. Epub 2012 Nov 16. PMID 23168366
- [Background] Van Cutsem E, Tabernero J, Lakomy R, Prenen H, Prausova J, Macarulla T, Ruff P, van Hazel GA, Moiseyenko V, Ferry D, McKendrick J, Polikoff J, Tellier A, Castan R, Allegra C. Addition of aflibercept to fluorouracil, leucovorin, and irinotecan improves survival in a phase III randomized trial in patients with metastatic colorectal cancer previously treated with an oxaliplatin-based regimen. J Clin Oncol. 2012 Oct 1;30(28):3499-506. doi: 10.1200/JCO.2012.42.8201. Epub 2012 Sep 4. PMID 22949147
- [Background] Tabernero J, Yoshino T, Cohn AL, Obermannova R, Bodoky G, Garcia-Carbonero R, Ciuleanu TE, Portnoy DC, Van Cutsem E, Grothey A, Prausova J, Garcia-Alfonso P, Yamazaki K, Clingan PR, Lonardi S, Kim TW, Simms L, Chang SC, Nasroulah F; RAISE Study Investigators. Ramucirumab versus placebo in combination with second-line FOLFIRI in patients with metastatic colorectal carcinoma that progressed during or after first-line therapy with bevacizumab, oxaliplatin, and a fluoropyrimidine (RAISE): a randomised, double-blind, multicentre, phase 3 study. Lancet Oncol. 2015 May;16(5):499-508. doi: 10.1016/S1470-2045(15)70127-0. Epub 2015 Apr 12. PMID 25877855
- [Background] Fuchs CS, Tomasek J, Yong CJ, Dumitru F, Passalacqua R, Goswami C, Safran H, Dos Santos LV, Aprile G, Ferry DR, Melichar B, Tehfe M, Topuzov E, Zalcberg JR, Chau I, Campbell W, Sivanandan C, Pikiel J, Koshiji M, Hsu Y, Liepa AM, Gao L, Schwartz JD, Tabernero J; REGARD Trial Investigators. Ramucirumab monotherapy for previously treated advanced gastric or gastro-oesophageal junction adenocarcinoma (REGARD): an international, randomised, multicentre, placebo-controlled, phase 3 trial. Lancet. 2014 Jan 4;383(9911):31-39. doi: 10.1016/S0140-6736(13)61719-5. Epub 2013 Oct 3. PMID 24094768
- [Background] Wilke H, Muro K, Van Cutsem E, Oh SC, Bodoky G, Shimada Y, Hironaka S, Sugimoto N, Lipatov O, Kim TY, Cunningham D, Rougier P, Komatsu Y, Ajani J, Emig M, Carlesi R, Ferry D, Chandrawansa K, Schwartz JD, Ohtsu A; RAINBOW Study Group. Ramucirumab plus paclitaxel versus placebo plus paclitaxel in patients with previously treated advanced gastric or gastro-oesophageal junction adenocarcinoma (RAINBOW): a double-blind, randomised phase 3 trial. Lancet Oncol. 2014 Oct;15(11):1224-35. doi: 10.1016/S1470-2045(14)70420-6. Epub 2014 Sep 17. PMID 25240821
- [Background] Garon EB, Ciuleanu TE, Arrieta O, Prabhash K, Syrigos KN, Goksel T, Park K, Gorbunova V, Kowalyszyn RD, Pikiel J, Czyzewicz G, Orlov SV, Lewanski CR, Thomas M, Bidoli P, Dakhil S, Gans S, Kim JH, Grigorescu A, Karaseva N, Reck M, Cappuzzo F, Alexandris E, Sashegyi A, Yurasov S, Perol M. Ramucirumab plus docetaxel versus placebo plus docetaxel for second-line treatment of stage IV non-small-cell lung cancer after disease progression on platinum-based therapy (REVEL): a multicentre, double-blind, randomised phase 3 trial. Lancet. 2014 Aug 23;384(9944):665-73. doi: 10.1016/S0140-6736(14)60845-X. Epub 2014 Jun 2. PMID 24933332